CLINICAL TRIAL: NCT04299984
Title: Italian Multicenter Prospective Database for Open Conversions and SemiConversions After Endovascular Aneurysm Repair
Brief Title: Italian Multicenter Database for Open Conversions After EVAR
Acronym: iConveRt
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Responsible Party: Principal Investigator, Paolo Perini, MD, PhD, Azienda Ospedaliero-Universitaria di Parma
Other Study IDs: iConveRt
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Abdominal Aortic Aneurysm; Abdominal Aortic Aneurysm Enlargement
Keywords: Abdominal aortic aneurysm; Open surgical conversion; Endovascular repair; EVAR explantation; Failed EVAR
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Open Conversions: Patients undergoing total or partial endograft explantation for any EVAR complication.
  Interventions: Procedure: Open Conversion after EVAR
- SemiConversions: Patients undergoing open or laparoscopic surgery for any EVAR complication (mostly endoleak correction) with complete endograft preservation.
  Interventions: Procedure: SemiConversion after EVAR

INTERVENTIONS:
Procedure: Open Conversion after EVAR — See "Open Conversions" group description.
  Groups: Open Conversions
Procedure: SemiConversion after EVAR — See "SemiConversions" group description.
  Groups: SemiConversions

SUMMARY:
Late endovascular abdominal aneurysm repair (EVAR) complications not amenable to endovascular correction can undergo either late open conversion (LOC) or semi-conversion (SC).

LOC is defined as a total or partial endograft explantation >30 days after the initial EVAR.

SC is defined as open or laparoscopic surgery for endoleak (EL) correction with complete endograft preservation.

The aim of this study is to collect in a prospective database the technical aspects of a multicenter experience of LOC and SC, and to analyse early and long-term outcomes of these two treatments.

ELIGIBILITY:
Inclusion Criteria:

* open or laparoscopic surgery for EVAR complications, with or without endograft explantation

Exclusion Criteria:

* endovascular reinterventions
* extra-anatomical bypass surgery (e.g. femoro-femoral crossover bypass) not associated with direct aorta/endograft surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent EVAR for abdominal aortic aneurysm exclusion, who developed complications not amenable to endovascular repair.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Early Mortality | 30 days
  30-day mortality after surgery
In-hospital Mortality | 90 days
  Mortality during in-hospital stay
Long-term survival | 4 years
  Long-term survival rate

SECONDARY OUTCOMES:
Early Morbidity | 30 days
  Major complications after surgery
Related complications | 4 years
  Aorta-related complications during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Perini, MD, Principal Investigator — Parma University Hospital
Locations (1):
- Azienda Ospedaliero-Universitaria di Parma, Parma, Italy

IPD SHARING:
Plan to Share IPD: No